CLINICAL TRIAL: NCT06844513
Title: HUGO RAS Robotic Platform for Radical Prostatectomy and Partial Nephrectomy: Comparison with the Da Vinci Robotic Platform
Brief Title: Comparison Between HUGO RAS Robotic Platform and Da Vinci Robotic Platform
Acronym: URO-ROBOT-2023
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URO ROBOT 2023
Record Dates: First submitted 2025-01-10; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer (Adenocarcinoma); Renal Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- prostate cancer (Active Comparator): Patients with prostate cancer (Group A), enrolled according to the inclusion criteria, are randomized to undergo radical prostatectomy (RP) using either the Da Vinci Xi platform (control group) or the HUGO™ RAS platform (study group).
  Interventions: Procedure: Radical prostatectomy
- kidney cancer (Active Comparator): patients with kidney cancer (Group B), enrolled according to the inclusion criteria, are randomized to undergo partial nephrectomy (PN) using either the Da Vinci Xi platform or the HUGO™ RAS platform.
  Interventions: Procedure: Partial nephrectomy

INTERVENTIONS:
Procedure: Radical prostatectomy — Radical prostatectomy performed using the Da Vinci Xi and the HUGO RAS platform
  Arms: prostate cancer
Procedure: Partial nephrectomy — partial nephrectomy (PN) using either the Da Vinci Xi platform or the HUGO™ RAS platform
  Arms: kidney cancer

SUMMARY:
The study is designed as a single-center, prospective, interventional, non-pharmacological, randomized, open-label, controlled trial with parallel groups. It targets patients with prostate cancer or kidney cancer who are candidates for robot-assisted surgical treatment, specifically radical prostatectomy (RP) or partial nephrectomy (PN).

DETAILED DESCRIPTION:
The study is designed as a single-center, prospective, interventional, non-pharmacological, randomized, open-label, controlled trial with parallel groups. It targets patients with prostate cancer or kidney cancer who are candidates for robot-assisted surgical treatment, specifically radical prostatectomy (RP) or partial nephrectomy (PN). The study is divided into a patient enrolment and robot-assisted treatment phase, followed by a phase of oncological and functional follow-up. Once enrolled, patients will be randomized to undergo treatment using either the Da Vinci Xi platform (Intuitive Surgical) or the HUGO™ RAS platform (Medtronic) according to block randomization.

Patients with prostate cancer (Group A), enrolled according to inclusion criteria, will be randomized to undergo RP treatment with the Da Vinci Xi platform (control group) or RP treatment with the HUGO™ RAS platform (study group).

Patients with kidney cancer (Group B), enrolled according to inclusion criteria, will be randomized to undergo PN treatment with the Da Vinci Xi platform or PN treatment with the HUGO™ RAS platform.

If the surgical, oncological, and functional outcomes observed following radical prostatectomy and partial nephrectomy performed with the HUGO RAS platform prove to be equivalent to those obtained with the Da Vinci Xi platform, it should lead to a progressive increase in the use of the HUGO RAS platform, resulting in a reduction in the overall costs associated with robotic urological surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients with Prostate Cancer (Group A)

* Age ≥ 18 years.
* Life expectancy greater than 10 years.
* Diagnosis of prostate cancer following prostate needle biopsy.
* Clinical stage cT1-T3b, N0-1 disease.
* Positive anesthetic fitness assessment for robot-assisted radical prostatectomy.
* Provision of informed consent for the study.

Patients with Kidney Cancer (Group B)

* Age ≥ 18 years.
* Radiological diagnosis of organ-confined kidney cancer at clinical stage T1a or T1b.
* Underwent CT and/or MRI of the abdomen with contrast medium.
* Positive anesthetic fitness assessment for robot-assisted partial nephrectomy.
* Provision of informed consent for the study.

Exclusion Criteria:

Patients with Prostate Cancer (Group A)

* Expression of a preference for radical treatment other than surgery (e.g., external radiotherapy).
* Metastatic prostate cancer (M1).
* Other conditions deemed by healthcare professionals to contraindicate inclusion in the study.

Patients with Kidney Cancer (Group B)

* Indication for radical nephrectomy.
* Metastatic kidney cancer (M1).
* Other conditions deemed by healthcare professionals to contraindicate inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2033-03-01 (Estimated)

PRIMARY OUTCOMES:
Equivalence of the HUGO RAS platform compared to the Da Vinci Xi robot in terms of perioperative complications | 90 days
  To demonstrate the equivalence of the HUGO RAS platform compared to the Da Vinci Xi robot in terms of perioperative complications observed within 90 days post-surgery. This evaluation will be conducted separately for:
  Patients undergoing radical prostatectomy (RP). Patients undergoing partial nephrectomy (PN).
  perioperative complication rate of grade greater than or equal to Clavien-Dindo IIIa within 90 days after surgery will be calculated.

SECONDARY OUTCOMES:
Equivalence between surgeries performed using the Da Vinci Xi and the HUGO RAS platform: Ergonomics for the primary and secondary operators | during surgery
Equivalence between surgeries performed using the Da Vinci Xi and the HUGO RAS platform: Operative times | during surgery
Equivalence between surgeries performed using the Da Vinci Xi and the HUGO RAS platform: Instrument conflicts or malfunctions | during surgery
  Instrument conflicts and malfunctions will be calculated (in number and %)
Equivalence between surgeries performed using the Da Vinci Xi and the HUGO RAS platform: Intraoperative blood loss | during surgery
Equivalence between surgeries performed using the Da Vinci Xi and the HUGO RAS platform: Length of hospital stay. | up to 4 days
Oncologic outcomes of PR or PN surgery - Rate of positive surgical margins | 90 days after surgery
Oncologic outcomes of PR or PN surgery : Survival time free of biochemical recurrence of disease. | 5 years
Oncologic outcomes of PR or PN surgery : - Metastasis-free survival time | 5 years
Oncologic outcomes of PR or PN surgery : Overall survival | 5 years
Oncologic outcomes of PR or PN surgery : Cancer-specific survival | 5 years
functional outcomes of PR or PN surgery: - International Index of Erectile Function (IIEF-5) score of recovery of sexual function | 5 years
  The possible scores for the IIEF-5 range from 5 to 25, and erectile dysfunction is classified into five categories based on the scores: severe (5-7), moderate (8-11), mild to moderate (12-16), mild (17-21), and no ED (22-25).
functional outcomes of PR or PN surgery: - Number of pads used | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Brunocilla, Prof, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy